CLINICAL TRIAL: NCT02020837
Title: A Pilot Study Assessing the Effect of Lymphaticovenous Micro-Anastomosis in the Treatment of Postmastectomy Lymphedema
Status: Terminated | Phase: Early Phase 1 | Type: Interventional
Why Stopped: Halted prematurely due to low enrollment
Sponsor: University of Arkansas (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 202676
Record Dates: First submitted 2013-12-19; First posted 2013-12-25 (Estimated); Results first posted 2018-04-09 (Actual); Last update posted 2018-06-27 (Actual); Status verified 2018-04

CONDITIONS: Lymphedema; Post Mastectomy
MeSH Terms: conditions — Lymphedema

STUDY DESIGN:
Intervention Model Description: A lymphatic diversion with lymphaticovenous microanastomosis will be performed.
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Lymphaticovenous Micro-Anastomosis (Experimental)
  Interventions: Procedure: Lymphaticovenous Micro-Anastomosis

INTERVENTIONS:
Procedure: Lymphaticovenous Micro-Anastomosis

SUMMARY:
This study will assess the impact of lymphaticovenous microanastomosis in volume reduction of postmastectomy upper extremity lymphedema. We hypothesize that multiple lymphaticovenous micro-anastomosis in the distal arm will result in the reduction of volume and improvement in quality of life of patients with post-mastectomy lymphedema

ELIGIBILITY:
Inclusion Criteria:

* Subject is 18-70 years of age
* Subject is Stage II-IV unilateral lymphedema

Exclusion Criteria:

* Subject is less than 6 months from completion of cancer treatment
* Subject has allergic reaction to the lymphatic contrast agent (Indocyanine Blue)
* Subject is medically unfit for the procedure
* Subject is unable to complete the follow-up visits
* Women with a positive urine pregnancy test are excluded from this study; women of childbearing potential (defined as those who have not undergone a hysterectomy or who have not been postmenopausal for at least 24 consecutive months) must agree to refrain from breast feeding and practice adequate contraception as specified in the informed consent. Adequate contraception consists of oral contraceptive, implantable contraceptives, injectable contraceptives, a double barrier method, or abstinence.
* Subject has bilateral lymphedema

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2014-09; Primary Completion 2015-12-03 (Actual); Study Completion 2017-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mauricio Moreno, MD, Principal Investigator — University of Arkansas
Locations (1):
- University of Arkansas for Medical Sciences, Little Rock, Arkansas, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Lymphaticovenous Micro-Anastomosis: Lymphaticovenous Micro-Anastomosis
Period: Overall Study
Arm/Group | Lymphaticovenous Micro-Anastomosis
Started | 2
Completed | 2
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Lymphaticovenous Micro-Anastomosis
Number analyzed (Participants) | 2
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 0
  >=65 years | 2
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 2
  More than one race | 0
  Unknown or Not Reported | 0
Count of Participants [Count of Participants; unit: Participants] — Number of participants
  Participants | 2

OUTCOME MEASURES:

1. Primary Outcome: Changes Relative to Baseline in the Volume of the Affected Limb at 3 and 6 Months From Surgery
Description: Lymphatic Volumetric Assessment. Evaluation of the volumetric change, relative to baseline measurement, in the volume of the affected limb at 3 and 6 months from the procedure.
Time Frame: 3 and 6 months from surgery
Population: Early termination leading to small numbers of subjects.Outcome measures not computed because data would not be statistically relevant.
Arm/Group | Lymphaticovenous Micro-Anastomosis
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | Lymphaticovenous Micro-Anastomosis
All-Cause Mortality (participants affected / at risk) | 0/2
Serious Adverse Events (participants affected / at risk) | 0/2
Other Adverse Events (participants affected / at risk) | 0/2

LIMITATIONS AND CAVEATS:
Early termination leading to small numbers of subjects. Outcome measures not computed because data would not be statistically relevant.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes